CLINICAL TRIAL: NCT05868564
Title: Determination Of Effectiveness Of Directional Atherectomy Followed By A Paclitaxel- Coated Balloon For The Treatment Of Infrainguinal Vessels With Long Occlusive Femoropopliteal Lesions
Brief Title: Atherectomy Followed With a Drug Coated Balloon in the Treatment of Long Femoropopliteal Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Second Affiliated Hospital of Soochow University (Other); Affiliated Hospital of Nantong University (Other); First Affiliated Hospital of Zhejiang University (Other); Zhejiang University (Other); Qingdao Hiser Medical Group (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The DEFINITIVE LL Study
Record Dates: First submitted 2023-03-07; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Atherectomy; drug coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atherectomy+Drug-coated balloon (Experimental): The lesion treated by atherectomy + UltrafreeTM drug-coated balloon.
  Interventions: Device: Atherectomy+Drug-coated balloon
- Drug-coated balloon (Active Comparator): The lesion treated by UltrafreeTM drug-coated balloon only.
  Interventions: Device: Drug-coated balloon

INTERVENTIONS:
Device: Atherectomy+Drug-coated balloon — Patients in experimental group will undergo endovascular treatment for femoropopliteal lesions. The lesion will be treated by atherectomy+drug-coated balloon in the experimental group
  Arms: Atherectomy+Drug-coated balloon
Device: Drug-coated balloon — drug-coated balloon only in the active comparator group.
  Arms: Drug-coated balloon

SUMMARY:
The study is a prospective, multicenter, randomized pilot study to evaluate the clinical outcome of the plaque atherectomy system followed by the UltrafreeTM drug coated balloon catheter versus the drug coated balloon in patients with chronic long femoropopliteal lesions.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, controlled comparison study. A total of 100 subjects will be enrolled into this study and will be randomized on a 1:1 basis to either drug coated balloon angioplasty combined with atherectomy or drug coated balloon angioplasty for subjects with long de-nove or restenosis femoropopliteal lesions( Stenotic lesion>15cm or Chronic total occlusion between 6-15cm). Angiographic patterns of the target lesion, including lesion length, calcification grade, and minimal lumen diameter (MLD) prior to and after the intervention, ultrasound images of the target lesion at 12-month follow-up will be independently adjudicated by an independent angiographic and ultrasound core lab. The primary endpoint is primary patency at 12 months based on Kaplan-Meier survival analysis. Follow-up visits are scheduled at 1,3,6,12,24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be between 18 and 85 years old;
2. Chronic, symptomatic lower limb ischemia defined as Rutherford categories 3-5;
3. Stenotic, restenosis, or occlusive lesions in the native femoropopliteal artery which meets all of the following criteria: Stenotic lesion(>70% diameter stenosis) >15cm or Chronic total occlusion between 6-15cm; Target vessel is 3.0 to 7.0 mm in diameter (visual estimate); Guidewire must be across the target lesion within the true lumen before study randomization;
4. Patent distal popliteal artery and at least one patent distal runoff;
5. Willing to comply with the follow-up evaluation;
6. Written informed consent prior to any study procedures.

Exclusion Criteria:

1. Women during pregnancy and lactation, or patients with baby planning;
2. Life expectancy<2 years;
3. Target lesion/vessel with in-stent restenosis
4. Target restenosis/vessel lesion previously treated with drug coated balloon or atherectomy <12 months
5. Subjects s who are currently participating in other interventional drug or device trials;
6. Angiographic evidence of thrombus within the target vessel
7. Subjects have a history of stroke within 3 months;
8. Subjects have a history of myocardial infarction, thrombolytic therapy, or angina pectoris within 2 weeks;
9. Concomitant Renal failure with a serum creatinine>2.0mg/dl; Subjects with known allergy to heparin, low molecular weight heparin, and contrast agents.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Peak Systolic Velocity Ratio (PSVR) | 12-month
  Peak Systolic Velocity Ratio (PSVR) of target lesion measured by ultrasound (PSVR ≤2.4 means primary patent of target lesion)
Freedom from major adverse limb events（MALEs） | 12-month
  Freedom from flow-limiting dissections (D-F), clinically-driven target vessel revascularization, major amputation, and all-cause of death

SECONDARY OUTCOMES:
Technical success | Immediately after endovascular treatment
  Defined as achievement of final residual diameter stenosis of <30% on the procedural completion angiogram, using the assigned device only, whereas lesion success is defined as achievement of <30% residual stenosis using any percutaneous method.
Procedural success | During the hospital stay
  Defined as technical or device success without the occurrence of major adverse events
Primary sustained clinical improvement | 24-month
  Defined as sustained upward shift of at least one category on the Rutherford classification without the need for repeated target lesion revascularization (TLR) in surviving patients
Quality of life score | 24-month
  Quality of Life (QOL) score at 24 months; The minimum value is 1, and the maximum value is 7. The higher scores mean a better outcome.
EuroQol five dimensions questionnaire (EQ 5D-5L) score | 24-month
  EQ 5D-5L score at 24 months；The minimum value is 0, and the maximum value is 5. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ye, M.D., Principal Investigator — Department of Vascular Surgery, Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China